CLINICAL TRIAL: NCT03683615
Title: Resorbable Polymer Plates in Repair of Blowout Orbital Floor Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Tamer Ismail Gawdat, clinical professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16111985
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Post-Traumatic Orbital Deformity
Keywords: Resorbable, blow out fractures
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with traumatic recent orbital blow out fractures (Other)
  Interventions: Procedure: repair of orbital floor fractures using resorbable plates

INTERVENTIONS:
Procedure: repair of orbital floor fractures using resorbable plates

SUMMARY:
It is a prospective study to evaluate the use of resorbable plates for the repair of blow out orbital floor fractures over a follow up period of one year at both cosmetic and functional levels.

ELIGIBILITY:
Inclusion Criteria:

* Class I, II blowout floor fracture.
* Presented within 2 weeks of trauma.
* Have muscle or soft tissue distortion with clinically significant diplopia, enophthalmos or restrictive strabismus.

Exclusion Criteria:

* Comminuted orbital fractures involving the rim.
* Associated globe injuries.
* Delayed presentation.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
anatomical reduction of the fracture | one month
  reduction of the fractured segment and restore the normal orbital volume and contents . assessment of reduction by measuring the changes in the orbital volume using computed tomography

SECONDARY OUTCOMES:
improvement of symptoms | 6 to 12 months
  improvement of the patient complaints as diplopia and enophthalmos using questionnaire